CLINICAL TRIAL: NCT04636541
Title: Goal Management Training Home-Based Approach for Cognitive Impairment in Parkinson's Disease: A Single-Blind Randomized Trial
Brief Title: Goal Management Training for Parkinson Disease Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AGiguère-Rancourt
Record Dates: First submitted 2020-10-30; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Parkinson Disease; Cognitive Intervention; Goal Management Training; Executive Functions
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Comparison of two different cognitive intervention (two groups, randomized, single blinded)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The research was a single blind randomized comparative study. After the screening evaluation, participants were randomly assigned to either group A or B, described below (block randomization, three blocks of four participants).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Management Training (Experimental): GMT modules were adapted for French-speaking patients with PD-MCI. Each session was reduced from nine 90-120-minute sessions (original GMT) to five 60-90-minute sessions, one session per week, in order to avoid fatigue. As for original GMT, participants were given exercises between sessions (mindfulness exercises and metacognitive reflections). In original-GMT, some information is repeated several times, but not in Adapted-GMT. Exercises demanding motor dexterity, such as card distribution, were removed. Adapted-GMT included information on PD-MCI and executive dysfunction (some psychoeducation). In addition, Adapted-GMT modules were administered individually with an iPad, as opposed to a power-point group presentation in original-GMT. A workbook was handed to participants, as in previous studies.
  Interventions: Behavioral: Goal Management Training
- Psychoeducation sessions coupled mindfulness exercises (Active Comparator): Five modules were designed as a discussion with patients and caregivers about various PD symptoms: module I-brain and motor symptoms; module II-autonomic symptoms; module III- psychological symptoms; module IV-brain and cognition; and module V-cognitive impairments in PD. Patients were handed the information book about the five modules at the beginning of the study. The objective was to improve their understanding of their condition and to discuss other components that could affect their cognitive abilities. After the 40-60-minute informative part, mindfulness exercises were offered for 20-30 minutes per session. Participants were not invited to practice exercises between sessions, but 3/6 participants reported they did.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Goal Management Training — Goal Management Training® (GMT) has been developed to improve executive functions. It was validated in patients presenting executive dysfunction following many conditions: acquired traumatic brain injury, neurodevelopmental spina bifida, attention deficit and hyperactivity disorder (ADHD), subjective cognitive complaints and multiple sclerosis. GMT includes self-instruction strategies, self-monitoring exercises, cognitive training techniques, psychoeducation on cognitive processes, mindfulness exercises and assignments between sessions. It has been shown to increase patient awareness of deficits and improve cognitive control in goal-directed behaviors. The original GMT is a nine-week program administered to dysexecutive patients in 90-to-120-minute group sessions. Thus, it might be suitable for PD-MCI patients presenting with executive dysfunction.
  Arms: Goal Management Training
Behavioral: Psychoeducation — See the Arm section for full details. For a justification of how we designed this intervention: Many clinical guidelines include general recommendations about giving information to PD patients and family so they can take part into decision process. However, few standardized psychoeducation interventions are available, and they don't include information on PD cognitive decline. Some studies investigated Mindfulness Based Stress Reduction (MBSR) and other related mindfulness interventions in PD patients. In this approach, formal meditative exercises are included to develop non-judgmental attention to experiences in the present moment. In elderly patients with MCI unrelated to PD, mindfulness interventions show positive effects on cognitive functioning, including attention, executive functioning and memory (Gard et al., 2014). Therefore, non-pharmacological interventions for PD-MCI including both education on cognitive symptoms, as well as mindfulness exercises, are promising.
  Arms: Psychoeducation sessions coupled mindfulness exercises

SUMMARY:
Mild cognitive impairment is experienced by approximately 30% of patients with Parkinson's disease (PD-MCI), often affecting executive functions. There is currently no pharmacological treatment available for PD-MCI and non-pharmacological treatments are still scarce. The aim of this study was to test preliminary efficacy/effectiveness of two home-based cognitive interventions adapted for patients with PD-MCI: Goal Management Training, adapted for PD-MCI (Adapted-GMT), and a psychoeducation program combined with mindfulness exercises. Twelve persons with PD-MCI with executive dysfunctions, as measured by extensive neuropsychological evaluation, were randomly assigned to one of two intervention groups. Both groups received five sessions each lasting 60-90 minutes for five weeks, in presence of the caregiver. Measures were collected at baseline, mid-point, at one-week, four-week and 12-week follow-ups. Primary outcomes were executive functions assessed by subjective (DEX questionnaire patient- and caregiver-rated) and objective (Zoo Map Test) measures. Secondary outcomes included quality of life (PDQ-39), global cognition (DRS-II), and neuropsychiatric symptoms (NPI-12). Safety data (fatigue, medication change and compliance) were also recorded. Repeated measures ANCOVAs were applied to outcomes. Both groups significantly ameliorated executive functions overtime as indicated by improvements in DEX-patient and DEX-caregiver scores. PDQ-39 scores decreased at the four-week follow-up in the Psychoeducation/Mindfulness group whereas they were maintained in the Adapted-GMT group. All other measures were maintained over time in both groups. Adapted-GMT and Psychoeducation/Mindfulness groups both improved executive functioning. This is one of the first studies to test home-based approaches, tailored to the participant's cognitive needs, and involving caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. PD diagnosis from the United Kingdom Research Brain Bank diagnostic criteria for PD (Hughes et al., 1992);
2. PD-MCI diagnosis from the Movement Disorder Society Task Force diagnostic criteria. Single and multiple-domain MCI were both included, only if executive functions were significantly impaired (-1 standard deviation on executive function tests according to age and education-adjusted norms);
3. Montreal Cognitive Assessment scores between 21 and 27;
4. Anti-Parkinson medication stable (at screening) since at least two months;
5. All other medications, including psychotropics, stable for at least three months.

Exclusion Criteria:

1. Participants with PD and dementia diagnosis
2. Patients with other neurological or psychiatric disorders.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Raw score Change from baseline DEX (self rated) to 3 weeks after beginning of intervention | 3 weeks after beginning of intervention (mid-point)
  Questionnaire on subjective executive functions
Raw score Change from baseline DEX (self rated) to 1 week post test | 1 week post-test
  Questionnaire on subjective executive functions
Raw score Change from baseline DEX (self rated) to 4 weeks post test | 4 weeks post-test
  Questionnaire on subjective executive functions
Raw score Change from baseline DEX (self rated) to 12 weeks post test | 12 weeks post-test
  Questionnaire on subjective executive functions
Raw score Change from baseline DEX (caregiver rated) to 3 weeks after the beginning of intervention | 3 weeks after beginning of intervention (mid-point)
  Questionnaire on subjective executive functions (caregiver rates the executive functions of the participant
Raw score Change from baseline DEX (caregiver rated) to 1 week post test | 1 week post-test
  Questionnaire on subjective executive functions (caregiver rates the executive functions of the participant
Raw score Change from baseline DEX (caregiver rated) to 4 weeks post test | 4 weeks post-test
  Questionnaire on subjective executive functions (caregiver rates the executive functions of the participant
Raw score Change from baseline DEX (caregiver rated) to 12 weeks post test | 12 weeks post-test
  Questionnaire on subjective executive functions (caregiver rates the executive functions of the participant
Raw score Change from baseline Zoo Map Test to 1 week post test | 1 week post-test
  Neuropsychological test assessing planification and organisation
Raw score Change from baseline Zoo Map Test to 4 weeks post test | 4 weeks post-test
  Neuropsychological test assessing planification and organisation
Raw score Change from baseline Zoo Map Test to 12 weeks post test | 12 weeks post-test
  Neuropsychological test assessing planification and organisation

SECONDARY OUTCOMES:
Raw score Change from baseline Parkinson Disease Questionnaire (39 items; PDQ-39) to 3 weeks after the beginning of intervention | 3 weeks after beginning of intervention (mid-point of intervention)
  Self rated questionnaire on quality of life with symptoms of Parkinson Disease
Raw score Change from baseline PDQ-39 to 1 week post-test | 1 week post-test
  Self rated questionnaire on quality of life with symptoms of Parkinson Disease
Raw score Change from baseline PDQ-39 to 4 weeks post-test | 4 weeks post-test
  Self rated questionnaire on quality of life with symptoms of Parkinson Disease
Raw score Change from baseline PDQ-39 to 12 weeks post-test | 12 weeks post-test
  Self rated questionnaire on quality of life with symptoms of Parkinson Disease
Mean Change from baseline Dementia Rating Scale, 2nd edition (DRS-II) to 1 week post-test | 1 week post-test
  A brief neuropsychological instrument designed to assess general cognitive functioning
Mean Change from baseline Dementia Rating Scale, 2nd edition (DRS-II) to 4 weeks post-test | 4 weeks post-test
  A brief neuropsychological instrument designed to assess general cognitive functioning
Mean Change from baseline Dementia Rating Scale, 2nd edition (DRS-II) to 12 weeks post-test | 12 weeks post-test
  A brief neuropsychological instrument designed to assess general cognitive functioning
Raw score Change from baseline Zarit Burden Interview (12 items) to 3 weeks after the beginning of intervention | 3 weeks after the beginning of intervention (mid-point)
  A 12-item questionnaire assessing the feeling of burden of the caregiver
Raw score Change from baseline Zarit Burden Interview (12 items) to 1 week post-test | 1 week post-test
  A 12-item questionnaire assessing the feeling of burden of the caregiver
Raw score Change from baseline Zarit Burden Interview (12 items) to 4 weeks post-test | 4 weeks post-test
  A 12-item questionnaire assessing the feeling of burden of the caregiver
Raw score Change from baseline Zarit Burden Interview (12 items) to 12 week post-test | Baseline, mid-point of intervention, 1 week post-test, 4 weeks post-test and 12 weeks post-test
  A 12-item questionnaire assessing the feeling of burden of the caregiver
Raw score Change from baseline Neuropsychiatric Inventory, 12 items to 3 weeks after the beginning of intervention (mid-point) | 3 weeks after the beginning of intervention (mid-point)
  assessment of twelve neuropsychiatric symptoms usually found in dementia
Raw score Change from baseline Neuropsychiatric Inventory, 12 items to 1 week post-test | 1 week post-test
  assessment of twelve neuropsychiatric symptoms usually found in dementia
Raw score Change from baseline Neuropsychiatric Inventory, 12 items to 4 weeks post-test | 4 week post-test
  assessment of twelve neuropsychiatric symptoms usually found in dementia
Raw score Change from baseline Neuropsychiatric Inventory, 12 items to 12 weeks post-test | 12 week post-test
  assessment of twelve neuropsychiatric symptoms usually found in dementia
Raw score Change from baseline Apathy Evaluation Scale (AES) to 3 weeks after the beginning of intervention (mid-point) | 3 weeks after the beginning of intervention (mid-point)
  An 18-item questionnaire assessing different aspects of apathy (cognitive, behavioral and emotional).
Raw score Change from baseline Apathy Evaluation Scale (AES) to 1 week post-test | 1 week post-test
  An 18-item questionnaire assessing different aspects of apathy (cognitive, behavioral and emotional).
Raw score Change from baseline Apathy Evaluation Scale (AES) to 4 weeks post-test | 4 weeks post-test
  An 18-item questionnaire assessing different aspects of apathy (cognitive, behavioral and emotional).
Raw score Change from baseline Apathy Evaluation Scale (AES) to 12 weeks post-test | 12 weeks post-test
  An 18-item questionnaire assessing different aspects of apathy (cognitive, behavioral and emotional).

CONTACTS AND LOCATIONS:
Overall Officials: Martine Simard, Study Director — Professor at Laval School of psychology
Locations (1):
- School of Psychology, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clare L, Teale JC, Toms G, Kudlicka A, Evans I, Abrahams S, Goldstein LH, Hindle JV, Ho AK, Jahanshahi M, Langdon D, Morris R, Snowden JS, Davies R, Markova I, Busse M, Thompson-Coon J. Cognitive rehabilitation, self-management, psychotherapeutic and caregiver support interventions in progressive neurodegenerative conditions: A scoping review. NeuroRehabilitation. 2018;43(4):443-471. doi: 10.3233/NRE-172353. PMID 30412509
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Dubois B, Burn D, Goetz C, Aarsland D, Brown RG, Broe GA, Dickson D, Duyckaerts C, Cummings J, Gauthier S, Korczyn A, Lees A, Levy R, Litvan I, Mizuno Y, McKeith IG, Olanow CW, Poewe W, Sampaio C, Tolosa E, Emre M. Diagnostic procedures for Parkinson's disease dementia: recommendations from the movement disorder society task force. Mov Disord. 2007 Dec;22(16):2314-24. doi: 10.1002/mds.21844. PMID 18098298
- [Background] Goldman JG, Vernaleo BA, Camicioli R, Dahodwala N, Dobkin RD, Ellis T, Galvin JE, Marras C, Edwards J, Fields J, Golden R, Karlawish J, Levin B, Shulman L, Smith G, Tangney C, Thomas CA, Troster AI, Uc EY, Coyan N, Ellman C, Ellman M, Hoffman C, Hoffman S, Simmonds D. Cognitive impairment in Parkinson's disease: a report from a multidisciplinary symposium on unmet needs and future directions to maintain cognitive health. NPJ Parkinsons Dis. 2018 Jun 26;4:19. doi: 10.1038/s41531-018-0055-3. eCollection 2018. PMID 29951580
- [Background] Grimes D, Gordon J, Snelgrove B, Lim-Carter I, Fon E, Martin W, Wieler M, Suchowersky O, Rajput A, Lafontaine AL, Stoessl J, Moro E, Schoffer K, Miyasaki J, Hobson D, Mahmoudi M, Fox S, Postuma R, Kumar H, Jog M; Canadian Nourological Sciences Federation. Canadian Guidelines on Parkinson's Disease. Can J Neurol Sci. 2012 Jul;39(4 Suppl 4):S1-30. doi: 10.1017/s031716710001516x. No abstract available. PMID 23126020
- [Background] Hindle JV, Watermeyer TJ, Roberts J, Brand A, Hoare Z, Martyr A, Clare L. Goal-orientated cognitive rehabilitation for dementias associated with Parkinson's disease-A pilot randomised controlled trial. Int J Geriatr Psychiatry. 2018 May;33(5):718-728. doi: 10.1002/gps.4845. Epub 2018 Jan 4. PMID 29314218
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Background] Jenkinson C, Peto V, Fitzpatrick R, Greenhall R, Hyman N. Self-reported functioning and well-being in patients with Parkinson's disease: comparison of the short-form health survey (SF-36) and the Parkinson's Disease Questionnaire (PDQ-39). Age Ageing. 1995 Nov;24(6):505-9. doi: 10.1093/ageing/24.6.505. PMID 8588541
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317
- [Background] Macht M, Gerlich C, Ellgring H, Schradi M, Rusinol AB, Crespo M, Prats A, Viemero V, Lankinen A, Bitti PE, Candini L, Spliethoff-Kamminga N, de Vreugd J, Simons G, Pasqualini MS, Thompson SB, Taba P, Krikmann U, Kanarik E. Patient education in Parkinson's disease: Formative evaluation of a standardized programme in seven European countries. Patient Educ Couns. 2007 Feb;65(2):245-52. doi: 10.1016/j.pec.2006.08.005. Epub 2006 Sep 11. PMID 16965885
- [Background] Matteau E, Dupre N, Langlois M, Provencher P, Simard M. Clinical validity of the Mattis Dementia Rating Scale-2 in Parkinson disease with MCI and dementia. J Geriatr Psychiatry Neurol. 2012 Jun;25(2):100-6. doi: 10.1177/0891988712445086. PMID 22689702
- [Background] Roy MA, Doiron M, Talon-Croteau J, Dupre N, Simard M. Effects of Antiparkinson Medication on Cognition in Parkinson's Disease: A Systematic Review. Can J Neurol Sci. 2018 Jul;45(4):375-404. doi: 10.1017/cjn.2018.21. Epub 2018 May 11. PMID 29747716
- [Background] Stamenova V, Levine B. Effectiveness of goal management training(R) in improving executive functions: A meta-analysis. Neuropsychol Rehabil. 2019 Dec;29(10):1569-1599. doi: 10.1080/09602011.2018.1438294. Epub 2018 Mar 14. PMID 29540124
- [Background] Vlagsma TT, Koerts J, Fasotti L, Tucha O, van Laar T, Dijkstra H, Spikman JM. Parkinson's patients' executive profile and goals they set for improvement: Why is cognitive rehabilitation not common practice? Neuropsychol Rehabil. 2016;26(2):216-35. doi: 10.1080/09602011.2015.1013138. Epub 2015 Feb 19. PMID 25693688
- [Background] Bora E, Walterfang M, Velakoulis D. Theory of mind in Parkinson's disease: A meta-analysis. Behav Brain Res. 2015 Oct 1;292:515-20. doi: 10.1016/j.bbr.2015.07.012. Epub 2015 Jul 9. PMID 26166188
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Marin RS, Biedrzycki RC, Firinciogullari S. Reliability and validity of the Apathy Evaluation Scale. Psychiatry Res. 1991 Aug;38(2):143-62. doi: 10.1016/0165-1781(91)90040-v. PMID 1754629
- [Background] Hiseman JP, Fackrell R. Caregiver Burden and the Nonmotor Symptoms of Parkinson's Disease. Int Rev Neurobiol. 2017;133:479-497. doi: 10.1016/bs.irn.2017.05.035. Epub 2017 Jul 21. PMID 28802929
- [Result] Couture M, Giguere-Rancourt A, Simard M. The impact of cognitive interventions on cognitive symptoms in idiopathic Parkinson's disease: a systematic review. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2019 Sep;26(5):637-659. doi: 10.1080/13825585.2018.1513450. Epub 2018 Sep 17. PMID 30221586
- [Result] Giguere-Rancourt A, Plourde M, Doiron M, Langlois M, Dupre N, Simard M. Goal management training (R) home-based approach for mild cognitive impairment in Parkinson's disease: a multiple baseline case report. Neurocase. 2018 Oct-Dec;24(5-6):276-286. doi: 10.1080/13554794.2019.1583345. Epub 2019 Mar 1. PMID 30821637
- [Derived] Giguere-Rancourt A, Plourde M, Racine E, Couture M, Langlois M, Dupre N, Simard M. Goal management training and psychoeducation / mindfulness for treatment of executive dysfunction in Parkinson's disease: A feasibility pilot trial. PLoS One. 2022 Feb 18;17(2):e0263108. doi: 10.1371/journal.pone.0263108. eCollection 2022. PMID 35180229